CLINICAL TRIAL: NCT02197208
Title: A Randomized Controlled Comparison of Spontaneous Natural Cycles and Human Chorionic Gonadotrophin-induced Natural Cycles in Frozen-thawed Embryos Transfer
Brief Title: A RCT Comparing Spontaneous Natural Cycles and Human Chorionic Gonadotrophin-induced Natural Cycles in FET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HKU-VL-NChCGFET
Record Dates: First submitted 2014-07-20; First posted 2014-07-22 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Subfertility; Pregnancy
Keywords: Frozen-thawed embryo transfer; natural cycle; spontaneous ovulation; hCG induced natural cycles
MeSH Terms: conditions — Infertility | interventions — Ultrasonography

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spontaneous NC (Active Comparator): Timing by the onset of LH surge as shown daily blood monitoring of serum estradiol and LH levels
  Interventions: Procedure: Daily monitoring of LH and E2; Device: ultrasound
- hCG induced NC (Experimental): Timing by giving hCG when the dominant follicle reaches >=17mm in diameter on ultrasound monitoring
  Interventions: Procedure: hCG induced natural cycle; Device: ultrasound

INTERVENTIONS:
Procedure: Daily monitoring of LH and E2 — ultrasound scanning would be carried out from 18 days before the expected period to confirm follicular growth, followed by daily blood monitoring of serum E2 and LH levels when the dominant follicle reaches 13-14mm in diameter. Ultrasound scanning can be arranged accordingly if the leading follicle remains less than 10mm in diameter. 5 ml of blood would be taken daily. LH surge is defined as the LH level being double of the average of the previous three days and higher than 20 IU/L. Ultrasound examination will be performed on the next day after the LH surge to measure the endometrial thickness. The transfer will be scheduled three or four days after the LH surge (for cleavage stage embryos) or six days after LH surge (for blastocyst transfer).
  Arms: Spontaneous NC
Procedure: hCG induced natural cycle — ultrasound monitoring would be started from 18 days before the expected period to monitor follicular growth, followed by USG every 2-3 days. hCG, 5,000-10,000 IU will be given when the leading follicle is >/= 17 mm and the endometrium measures >/=8 mm. Serum E2, LH and progesterone levels will be measured on the day of hCG. Embryo transfer would be scheduled on the fourth or fifth days after hCG injection (for cleavage stage embryos) or seventh days (for blastocyst transfer).
  Arms: hCG induced NC
Device: ultrasound

SUMMARY:
This is a randomized controlled trial on the comparison of the ongoing pregnancy rate in frozen-thawed embryo transfer cycles with spontaneous ovulation and hCG-induced natural cycles.

DETAILED DESCRIPTION:
Embryo cryopreservation is essential nowadays. It allows the usage of surplus good quality embryos in frozen-thawed embryo transfer (FET) cycles which avoids embryo wastage and facilitates the adoption of transferring a small number of embryos in the fresh stimulation cycle so as to reduce the risk of multiple pregnancy during in vitro fertilization (IVF) treatment. Elective cryopreservation of all fresh embryos is also required in special circumstances where fresh transfer is undesirable, for example in cases where a high risk of ovarian hyperstimulation syndrome is anticipated. Fresh transfer is not advisable when serum progesterone level is elevated or hydrosalpinx is detected during ovarian stimulation.

The availability of FETs would increase the likelihood of successful pregnancy from a single superovulation and oocyte retrieval cycle. It has been estimated that in modern IVF programmes which incorporates embryo cryopreservation, up to 42% of all conceptions could be derived from FET (Borini et al, 2008).

Although the pregnancy rate in FET is comparable with stimulated IVF cycles, the optimal regimen to prepare the endometrium for implantation is not yet well proven. By a recent Cochrane review, there is no evidence to prove the use of one regimen in preference to another (Ghobara T 2008).

Natural cycles (NC) are considered the best regimen as it is physiological, where natural conception occurs in. However, there are two most commonly employed methods to time the ovulation in natural cycles. One is to use ultrasound (USG) to monitor the follicular growth and endometrial thickness, with the use of human chorionic gonadotrophin (hCG) to trigger ovulation in the presence of a dominant follicle around 17-18mm in diameter. Another is to monitor the blood hormonal concentration to detect the luteinising hormone (LH) surge associated with natural ovulation. There is scarce information in this area as only one randomized controlled trial compared these two approaches. The authors aimed to recruit 240 subjects, but the study was prematurely terminated as significant results were resulted in the first interim analysis when the sample size reached 124. The ongoing pregnancy rate was 31.1% in the group with spontaneous LH surge and 14.3% in the hCG-induced group (Fatemi et al., 2010).

The use of natural LH surge and hCG trigger in intrauterine insemination was compared too. A meta-analysis revealed a significantly higher clinical pregnancy rate in IUI cycles with natural LH surge than that with hCG trigger. However, the data from randomized controlled trial showed no significant difference. Also the data were contradictory when the analysis confined to a specific indication of subfertility (Kosmas et al., 2007). A cochrane review in 2012 also suggested there was no evidence to advise that any regimen was better than another (Cantineau et al., 2012).

This randomized controlled trial aims to compare the ongoing pregnancy rate of FET in spontaneous NC and hCG-induced NC. The hypothesis of this trial is that the ongoing pregnancy rate of FET is similar for spontaneous NC and hCG-induced NC. The advantage of hCG-induced NC is likely a reduction in the duration of monitoring for timing FET when compared with spontaneous NC.

ELIGIBILITY:
Inclusion Criteria:

* Age of women <43 years
* Regular menstrual cycles ranging from 21-35 days with not more than 4 days variation between cycles
* Undergoing FET in natural cycles
* Normal uterine cavity as shown on saline sonogram performed before the IVF cycle or normal uterine cavity shown on pelvic scanning during the stimulated IVF cycle
* Endometrial thickness >=8mm in both stimulated IVF and FET cycles

Exclusion Criteria:

* >3 previous IVF cycles
* >6 embryos replaced without pregnancy
* Irregular menstrual cycles
* Subjects requiring clomid-induced cycles and hormonal replacement (HRT) cycles
* History of previous FET cycles within the study period
* Blastocyst transfer
* Preimplantation genetic diagnosis treatment
* Use of donor oocytes
* Presence of hydrosalpinx not corrected surgically prior to FET
* Recurrent miscarriage
* Serum progesterone level on the day of LH surge or day of hCG >5 nmol/L or 1.5 pg/L (these patients will be retrospectively excluded)
* Refusal to join the study

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2014-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
ongoing pregnancy rate | 12 weeks after embryos transfer
  the ongoing pregnancy rate which is defined as the number of viable pregnancies beyond 10-12 weeks gestation per transfer cycle

SECONDARY OUTCOMES:
Days of monitoring for timing FET | 4 weeks after last menstrual period
  The number of days needed for the monitoring for the timing of FET
Endometrial thickness on day of hCG or the next day after LH surge | 2-3 weeks after LMP
  The measurement of the endometrial thickness on the day of hCG or the next day after LH surge
Implantation rate | 4-6 weeks after embryo transfer
  Implantation rate: number of gestational sacs per number of embryos transferred
pregnancy rate | 2-4 weeks after embryo transfer
  number of positive pregnancy rate per transfer
Clinical pregnancy rate | 6-8 weeks after embryo transfer
  Number of pregnancy with positive fetal pulsation on scanning at 6 weeks of gestation.
Miscarriage rate | 20 weeks after embryo transfer
  rate of pregnancy loss <20 weeks per transfer cycles
Multiple pregnancy rate | 20 weeks after embryo transfer
  The rate of multiple pregnancy after ET

CONTACTS AND LOCATIONS:
Overall Officials: Vivian CY Lee, MBBS, Principal Investigator — Queen Mary Hospital / University of Hong Kong.
Locations (2):
- Center for Reproductive Medicine, Department of Obstetrics and Gynecology, Nanfang Hospital, Southern Medical University, Guangzhou, China
- Queen Mary Hospital, Hong Kong, Hong Kong, Hong Kong